

#### TRIAL STATISTICAL ANALYSIS PLAN

Document No.: c41671420-01

BI Trial No.: 1305-0024

**Title:** Pharmacokinetics, safety and tolerability of doses of BI 1015550

in healthy Chinese male and female subjects (open-label, parallel

group design)

(including Protocol Amendment No.1 [c39429830-02]).

Investigational

**Product:** 

BI 1015550

Responsible trial statistician:



Date of statistical

20 JUN 2023 SIGNED

analysis plan:

Version: 1

**** 

#### Proprietary confidential information

© 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies. All rights reserved. This document may not - in full or in part - be passed on, reproduced, published or otherwise used without prior written permission.

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.

# 1. TABLE OF CONTENTS

Date: 13 JUN 2023, Version 1.0

| TITLE | PAGE | 1 |
|--------------|------------------------------------------------|----|
| 1. | TABLE OF CONTENTS | 2 |
| 2. | LIST OF ABBREVIATIONS | |
| 3. | INTRODUCTION | 6 |
| <b>5.</b> | ENDPOINTS | |
| <b>5.1</b> | PRIMARY ENDPOINTS | |
| <b>5.2</b> | SECONDARY ENDPOINTS | |
| <b>5.2.1</b> | Key secondary endpoints | |
| 5.2.2 | Secondary endpoint | |
| 5.3 | FURTHER ENDPOINTS | 8 |
| <b>6.</b> | GENERAL ANALYSIS DEFINITIONS | |
| 6.1 | TREATMENTS | |
| 6.2 | IMPORTANT PROTOCOL DEVIATIONS | |
| 6.3 | INTERCURRENT EVENTS | |
| 6.4 | SUBJECT SETS ANALYSED | |
| 6.6 | HANDLING OF MISSING DATA AND OUTLIERS | 13 |
| 6.7 | BASELINE, TIME WINDOWS AND CALCULATED VISITS | |
| | PLANNED ANALYSIS | |
| 7.<br>7.1 | DEMOGRAPHIC AND OTHER BASELINE CHARACTERISTICS | |
| 7.1<br>7.2 | CONCOMITANT DISEASES AND MEDICATION | |
| 7.3 | TREATMENT COMPLIANCE | |
| 7.4 | PRIMARY OBJECTIVE ANALYSIS | |
| 7.4.1 | Main analysis | |
| 7.5 | SECONDARY OBJECTIVE ANALYSIS | |
| 7.5.1 | Key secondary objective analysis | |
| 7.5.2 | Secondary objective analysis | |
| 7.6<br>7.7 | FURTHER OBJECTIVE ANALYSIS EXTENT OF EXPOSURE | |
| 7.7<br>7.8 | SAFETY ANALYSIS | |
| 7.8.1 | Adverse Events | |
| 7.8.2 | Laboratory data | |
| 7.8.3 | Vital signs | |
| 7.8.4 | ECG | |
| 7.9 | OTHER ANALYSIS | |
| <b>7.9.1</b> | Biomarker analyses | |
| 7.9.2 | PK/PD analyses | 22 |

# Boehringer Ingelheim TRIAL STATISTICAL ANALYSIS PLAN 1305-0024


| 05-0024 | c41671420-01 |
|---|---|
| Proprietary confidential information © 2023 Boehringer Ingelheim In | nternational GmbH or one or more of its affiliated companies. |

| F10 | prictary confidential information © 2023 Bochringer ingenienti international Oniori of one of more of its armiated compa | illes. |
|---|---|---|
| 8. | TIMEPOINT OF RELEASE OF TREATMENT INFORMATION | 23 |
| 9. | REFERENCES | 24 |
| 11. | HISTORY TABLE | 27 |

# Boehringer Ingelheim TRIAL STATISTICAL ANALYSIS PLAN 1305-0024

**** 

c41671420-01

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.

## LIST OF TABLES

| Table 6.1: 1 | Treatments and labels used in the analysis | 1 | ( |
|--------------|--------------------------------------------|---|---|
| | Subject sets analysed | | |
| | History table | | |

Date: 13 JUN 2023, Version 1.0 BI-VQD-12681\_50-415\_AD-01 (4.0)

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.

# 2. LIST OF ABBREVIATIONS

See Medicine Glossary:


http://glossary

| Term | Definition / description |
|---|---|
| ALT | Alanine Aminotransferase |
| AST | Aspartate Aminotransferase |
| $\mathrm{AUC}_{0\text{-}\infty}$ | Area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity |
| BMI | Body mass index |
| $C_{\text{max}}$ | Maximum measured concentration of the analyte in plasma |
| CTP | Clinical trial protocol |
| CTR | Clinical trial report |
| CV | Arithmetic Coefficient of Variation |
| DILI | Drug induced liver injury |
| gCV | Geometric Coefficient of Variation |
| gMean | Geometric Mean |
| Max | Maximum |
| Min | Minimum |
| N | Number non-missing observations |
| P10 | 10th percentile |
| P90 | 90th percentile |
| PKS | PK parameter analysis set |
| Q1 | 1st quartile |
| Q3 | 3rd quartile |
| RPM | Report Planning Meeting |
| RAGe | Report Appendix Generator system |
| SD | Standard Deviation |
| TS | Treated Set |
| TSAP | Trial Statistical Analysis Plan |
| ULN | Upper Limit of Normal |

**** 

c41671420-01

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.

#### 3. INTRODUCTION


As per ICH E9  $(\underline{1})$ , the purpose of this document is to provide a more technical and detailed elaboration of the principal features of the analysis described in the protocol, and to include detailed procedures for executing the statistical analysis of the primary and secondary variables and other data.

This trial statistical analysis plan (TSAP) assumes familiarity with the Clinical Trial Protocol (CTP), including Protocol Amendments. In particular, the TSAP is based on the planned analysis specification as written in CTP Section 7 "Statistical Methods and Determination of Sample Size". Therefore, TSAP readers may consult the CTP for more background information on the study, e.g., on study objectives, study design and population, treatments, definition of measurements and variables, planning of sample size, randomization.

Study data (including data entered in the RAVE EDC system and external data provided by suppliers) will be stored in a Clinical Data Repository (CDR).

| Pharmacokinetic (PK) parameters will be ca<br>(version 8.1.1 or higher,<br>version). | alculated using Phoenix WinNonlin <sup>TM</sup> software ) or SAS Version 9.4 (or later |
|---|---|
| The statistical analyses will be performed wincluding SAS <sup>TM</sup> (current Version 9.4, by of SAS <sup>TM</sup> -based tools (e.g., macros for the a | ithin the validated working environment CARE, ), and a number analyses of AE data or laboratory data; Report impilation/formatting of the CTR appendices). |

# Boehringer Ingelheim TRIAL STATISTICAL ANALYSIS PLAN 1305-0024

**** 

c41671420-01

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.

Date: 13 JUN 2023, Version 1.0 BI-VQD-12681\_50-415\_AD-01 (4.0)

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.

#### 5. ENDPOINTS

#### 5.1 PRIMARY ENDPOINTS

#### **Section 2.1.2 of the CTP:**

The following pharmacokinetic parameters will be determined for BI 1015550:

- $AUC_{0-\infty}$  (area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity)
- $C_{max}$  (maximum measured concentration of the analyte in plasma)

#### 5.2 SECONDARY ENDPOINTS

# 5.2.1 Key secondary endpoints

This section is not applicable as no key secondary endpoints have been defined in the CTP.

#### 5.2.2 Secondary endpoint

#### Section 2.1.3 of the CTP:

The occurrence of any treatment-emergent adverse events, assessed as the percentage of subjects treated with investigational drug who experience such an event.

#### 5.3 FURTHER ENDPOINTS

#### Safety and tolerability endpoints

#### Section 2.2.2.1 of the CTP:

Safety and tolerability of BI 1015550 will be assessed based on:

- AEs (including clinically relevant findings from the physical examination)
- Safety laboratory tests
- 12-lead ECG


• Vital signs (blood pressure [BP], pulse rate [PR])




c41671420-01

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.



Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.

#### 6. GENERAL ANALYSIS DEFINITIONS

#### 6.1 TREATMENTS

For basic study information on treatments to be administered, assignment of treatment groups, selection of doses, refer to CTP Sections 3 and 4.

This trial is designed as open-label, single-dose with parallel dose groups.

It is planned to include a total of 24 healthy Chinese male and female subjects in the trial (12 subjects sequentially allocated to one of two ascending dose groups, with at least 3 female subjects within each dose group).

For details of dosage and formulation see Table 6.1:1 below.

Table 6.1: 1 Treatments and labels used in the analysis

| Tr | eatment | Short label |
|----|-------------------------------------------------------|-------------|
| A | BI 1015550 9 mg, TABLET, FILM COATED ONCE ORAL 9 mg | BI 9mg |
| В | BI 1015550 18 mg, TABLET, FILM COATED ONCE ORAL 18 mg | BI 18mg |

#### Section 1.2.2 of the CTP:

The Residual Effect Period (REP) of BI 1015550 is 7 days. This is the period after the last dose with measurable drug levels and / or pharmacodynamic effects still likely to be present.

Based on this, the following study phases will be defined for the analysis of adverse events (AEs):

### Screening

- Ranging from 0:00h on day of informed consent until time of first drug administration.
- On treatment (labelled with short label "BI 9mg", "BI 18mg")
  - o Ranging from the time of respective drug administration until 7 days (168 h) thereafter OR until trial termination (0:00 h on the day after trial termination), whatever occurs first.
- Follow-up (labelled "F/U")
  - Ranging from the end of REP until trial termination (0:00 h on the day after trial termination).

#### **Section 7.2.5 of the CTP:**

Note that AEs occurring after the last per protocol contact but entered before data base lock will be reported to Pharmacovigilance only and will not be captured in the trial database.


c41671420-01

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.

The following AE displays will be provided in the report:

In Section 15.3 and Appendix 16.1.13.1.8 (for ClinicalTrials.gov only) of the CTR displays, the on treatment phase will be analysed (labelled with the short label of the study treatment). The screening and follow-up phases will not be included in this analysis.

The following totals will be provided in addition for Section 15.3:

• a total over all BI treated on treatment phases ("BI Total")

In Section 15.4 and Appendix 16.2 (Listings) of the CTR displays, the screening period, as well as the follow-up phases will additionally be included and no totals will be provided.

For detailed information on the handling of the treatments refer to Technical TSAP ADS (analysis data set) plan and Analysis Data Reviewers guide.

#### 6.2 IMPORTANT PROTOCOL DEVIATIONS

Data discrepancies and deviations from the CTP will be identified for all treated subjects. Consistency check listings (for identification of deviations of time windows) and a list of protocol deviations (e.g. deviations in drug administration, in blood sampling times, etc.) will be provided to be discussed at the Report Planning Meeting (RPM). At this meeting, all manual deviations identified at the sites by the CRAs and deviations too complex to program will be reviewed by the trial team to decide which are considered important. For definition of important protocol deviations (iPD), and for the process of identification of these, refer to the Boehringer Ingelheim (BI) SOP "Identify and Manage Important Protocol Deviations (iPD)" (2).

Important protocol deviation (iPD) categories are pre-specified in the iPD specification file (DV domain) (3). IPDs will be identified no later than in the Report Planning Meeting, and the iPD categories will be updated as needed.

If any iPDs are identified, they are to be summarised into categories and will be captured in the iPD specification file (DV domain) (3) and in the decision log (4). Both documents will be stored within the TMF in EDMS.

The iPDs will be summarized and listed in the CTR.

#### 6.3 INTERCURRENT EVENTS

This section is not applicable.


Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.

#### 6.4 SUBJECT SETS ANALYSED

#### Section 7.2.1.1 of the CTP:

Statistical analyses will be based on the following analysis sets:

- Treated set (TS): The treated set includes all subjects who were treated with at least one dose of trial drug. The treated set will be used for safety analyses.
- Pharmacokinetic parameter analysis set (PKS): This set includes all subjects in the treated set (TS) who provide at least one PK endpoint that was defined as primary and was not excluded due to a protocol deviation relevant to the evaluation of PK or due to PK non-evaluability (as specified in CTP Section 7.2.1.2 and below). Thus, a subject will be included in the PKS, even if he/she contributes only one PK parameter value to the statistical assessment. Descriptive analyses of PK parameters will be based on the PKS.

The pharmacokinetic parameters listed in CTP Section 2.1 and 2.2.2 for drug BI 1015550, R-BI 1015550 and S-BI 1015550 will be calculated according to the relevant BI internal procedures.

Plasma concentration data and parameters of a subject will be included in the statistical pharmacokinetic (PK) analyses if they are not flagged for exclusion due to a protocol deviation relevant to the evaluation of PK (to be decided no later than in the Report Planning Meeting) or due to PK non-evaluability (as revealed during data analysis, based on the criteria specified below). Exclusion of a subject's data will be documented in the CTR.

Important protocol deviations may be

- Incorrect trial medication taken, i.e. the subject received at least one dose of trial medication the subject was not assigned to
- Incorrect dose of trial medication taken
- Use of restricted medications


Plasma concentrations and/or parameters of a subject will be considered as non-evaluable, if for example

- The subject experienced emesis that occurred at or before two times median t<sub>max</sub> of the respective treatment (Median t<sub>max</sub> is to be determined excluding the subjects experiencing emesis),
- Missing samples/concentration data at important phases of PK disposition curve

Plasma concentration data and parameters of a subject which are flagged for exclusion will be reported with its individual values but will not be included in the statistical analyses.

Only concentration values within the validated concentration range and actual sampling times will be used for the calculation of pharmacokinetic parameters. Concentrations used in the pharmacokinetic calculations will be in the same format provided in the bioanalytical report, (that is, to the same number of decimal places provided in the bioanalytical report).

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.

Table 6.4: 1 Subject sets analysed

| | Subject set | |
|----------------------------------|-------------|-----|
| Class of analysis | TS | PKS |
| Primary and further PK endpoints | | X |
| Safety & treatment exposure | X | |
| Demographic & baseline | X | |



#### 6.6 HANDLING OF MISSING DATA AND OUTLIERS

Handling of missing data and outliers will be performed as described in the CTP, Section 7.3:

Missing or incomplete AE dates are imputed according to BI standards (see BI-KMED-BDS-

Missing or incomplete AE dates are imputed according to BI standards (see BI-KMED-BDS-HTG-0035)  $(\underline{5})$ .

Missing data and outliers of PK data are handled according to BI standards. PK parameters that cannot be reasonably calculated based on the available drug concentration-time data will not be imputed.

#### 6.7 BASELINE, TIME WINDOWS AND CALCULATED VISITS

The baseline value is defined as the last measurement before trial drug administration.

#### **Section 6.1 of the CTP:**


Exact times of measurements outside the permitted time windows will be documented. The acceptable time windows for screening and the end of trial examination are provided in the CTP Flow Chart.

Trial measurements and assessments scheduled to occur 'before' trial medication administration on Day 1 are to be performed and completed within a 3 h-period prior to the trial drug administration.

The acceptable deviation from the scheduled time for vital signs, ECG, laboratory tests, and AEs/concomitant therapies questioning will be:

 $\pm$  30 min up to 48 h after drug administration (planned time)

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.

#### $\pm$ 120 min after 48 h to the end of study


If several activities are scheduled at the same time point in the Flow Chart, ECG should be the first and meal the last activity. Furthermore, if several measurements including venipuncture are scheduled for the same time, venipuncture should be the last of the measurements due to its inconvenience to the subject and possible influence on physiological parameters.

For planned blood sampling times, refer to the CTP Flow Chart. While these nominal times should be adhered to as closely as possible, the actual sampling times will be recorded and used for the determination of pharmacokinetic parameters.

Adherence to time windows will be checked via the consistency check listings at the RPM.

Unscheduled measurements of laboratory data and vital signs data will be assumed to be repeat measurements of the most recent scheduled measurement (e.g. for follow-up or confirmation of a particular value). Therefore, unscheduled measurements will be assigned to the planned time point of the previous scheduled measurement.

BI-VQD-12681\_50-415\_AD-01 (4.0)


c41671420-01

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.

#### 7. PLANNED ANALYSIS

Safety analysis (refer to Section 7.8) will be performed by will be presented in Sections 15.1 to 15.4 of the CTR and in Appendix 16.2 and 16.1.13.1.

Descriptive data analysis of PK endpoints and concentrations will be performed by the at BI and will be presented in Section 15.6 of the CTR and in Appendix 16.1.13.5.

The format of the listings and tables will follow the BI standards (see "Standards for Reporting of Clinical Trials and Project Summaries" (8)) with the exception of those generated for PK-calculations following BI standards for PK/PD analysis (9).

The individual values of all subjects will be listed, sorted by treatment group, subject number and visit. The listings will be included in Appendix 16.2 of the CTR.

The following standard descriptive statistical parameters will be displayed in summary tables of continuous variables:

N number non-missing observations

Mean arithmetic mean SD standard deviation

Min minimum Median median Max maximum

For analyte concentrations and PK parameters, the following descriptive statistics will additionally be calculated:

Nobs number of observations

CV arithmetic coefficient of variation

gMean geometric mean

gCV geometric coefficient of variation

P10 10<sup>th</sup> percentile Q1 1<sup>st</sup> quartile Q3 3<sup>rd</sup> quartile P90 90<sup>th</sup> percentile


The data format for descriptive statistics of concentrations will be identical to the data format of the respective concentrations. The descriptive statistics of PK parameters will be calculated using the individual values with the number of decimal places as provided by the evaluation program. Then the individual values as well as the descriptive statistics will be reported with three significant digits in the CTR.

Tabulations of frequencies for categorical data will include all possible categories available in the CRF and will display the number of observations in a category, as well as the percentage (%). Percentages will be rounded to one decimal place and will be based on all subjects in the

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.

respective subject set whether they have non-missing values or not. The category 'missing' will be displayed only if there are actually missing values.

Units of variables should be given in the titles or column/row descriptors in brackets (e.g. (mg)).

#### Exclusion of PK parameters

The ADS "ADPP" (PK parameters) contains column variables APEX and APEXCO indicating inclusion/exclusion (APEX) of a PK parameter and an analysis flag comment (APEXCO). All analyses based on the PKS will include parameters only if they are not flagged for exclusion, that is APEX is equal to "Included".

#### Exclusion of PK concentrations


The ADS "ADPC" (PK concentrations per time-point or per time-interval) contains column variables ACEX and ACEXCO indicating inclusion/exclusion (ACEX) of a concentration and an analysis flag comment (ACEXCO). Exclusion of a concentration depends on the analysis flag comment ACEXCO. For example, if ACEXCO is set to

- 'ALL CALC', the value will be excluded for all types of analyses based on concentrations.
- 'DESC STATS' the value will be excluded from descriptive evaluations per planned time point/time interval.
- to 'HALF LIFE', the value will be excluded from half-life calculation (and, as a consequence, any calculation that relies on  $\lambda_z$ ) only; the value is included for all other analyses.

If ACEXCO contains the addition 'TIME VIOLATION' or 'TIME DEVIATION' the value can be used for further analyses based on actual times. Excluded concentration itself will be listed in the CTR associated with an appropriate flag.

Further details are given in "Noncompartmental Pharmacokinetic / Pharmacodynamic Analyses of Clinical Studies" (7) and "Description of Analytical Transfer Files and PK/PD Data Files" (10).

#### 7.1 DEMOGRAPHIC AND OTHER BASELINE CHARACTERISTICS

Only descriptive statistics are planned for this section of the report, based on the TS. The data will be summarised by treatment group and in total.

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.

#### 7.2 CONCOMITANT DISEASES AND MEDICATION

Only descriptive statistics are planned for this section of the report, based on the TS.

Concomitant diseases and non-drug therapies will be coded according to the version defined in the decision log (4) of the coding system of the Medical Dictionary for Drug Regulatory Activities (MedDRA). Concomitant medications will be coded according to the most recent version of the World Health Organization Drug Dictionary (WHO-DD). The coding version number will be displayed as a footnote in the respective output.

#### Section 7.2.5 of the CTP:

Previous and concomitant therapies will be presented per treatment group without consideration of time intervals and treatment periods.

The diagnoses and medications will be listed. Subjects without any concomitant diagnoses or concomitant therapies will be marked with a "No" in the respective column.

The relevance of the concomitant therapies to the evaluation of PK data will be decided no later than at the RPM.

#### 7.3 TREATMENT COMPLIANCE

#### Section 4.3 of the CTP:

Compliance will be assured by administration of all trial medication in the trial centre under supervision of the investigating physician or a designee. The measured plasma concentrations of trial medication will provide additional confirmation of compliance.

It is not intended to list the compliance separately. Any deviations from complete intake will be addressed in the RPM and described in the CTR.

#### 7.4 PRIMARY OBJECTIVE ANALYSIS

#### 7.4.1 Main analysis

#### Section 7.2.2 of the CTP:


The primary endpoints (refer to Section 5.1) will be calculated according to BI standards. The analysis will be based on the PKS and will be descriptive in nature.



Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.



#### 7.5 SECONDARY OBJECTIVE ANALYSIS

#### 7.5.1 Key secondary objective analysis

This section is not applicable as no key secondary endpoint has been specified in the protocol.

#### 7.5.2 Secondary objective analysis

The analysis of secondary safety endpoint will be based on the TS and will be descriptive in nature (refer to Section 7.8).

#### 7.6 FURTHER OBJECTIVE ANALYSIS



#### Safety endpoints

For a description of the analysis of safety and tolerability, please refer to Section 7.8.

#### 7.7 EXTENT OF EXPOSURE

Descriptive statistics are planned for this section of the report based on the TS. The date and time of drug administration will be listed for each subject.

#### 7.8 SAFETY ANALYSIS

All safety analyses will be performed on the TS.

The safety data for treated subjects who failed to complete the study (dropouts or withdrawals) will be reported as far as their data are available. All withdrawals will be documented and the reason for withdrawal recorded.

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.

#### 7.8.1 Adverse Events

AEs will be coded using MedDRA. The coding version number will be displayed as a footnote in the respective output.

Unless otherwise specified, the analyses of AEs will be descriptive in nature. All analyses of AEs will be based on the number of subjects with AEs and NOT on the number of AEs. BI standards as presented in "Analysis and Presentation of Adverse Event Data from Clinical Trials – Display Template" (11) and "Analysis and Presentation of AE data from clinical trials" (12) will be applied.

The analysis of AEs will be based on the concept of treatment emergent AEs. That means that all AEs will be assigned to 'screening', 'on-treatment' or 'follow-up' phases as defined in Section 6.1. AEs will be analysed based on actual treatments, as defined in Table 6.1: 1.

According to the clinical study protocol, adverse events of special interest (AESI) will be analysed:

#### Section 5.2.6.1.4 of the CTP:

The following are considered as AESIs:

#### • Potential severe DILI


A potential severe Drug Induced Liver Injury (DILI) that requires follow-up is defined by the following alterations of hepatic laboratory parameters:

- o An elevation of AST (aspartate aminotransferase) and/or ALT (alanine aminotransferase)  $\geq$ 3-fold ULN combined with an elevation of total bilirubin  $\geq$ 2-fold ULN measured in the same blood sample, or in samples drawn within 30 days of each other, or
- o Aminotransferase (ALT, and/or AST) elevations  $\geq$ 10-fold ULN

These lab findings constitute a hepatic injury alert and the subjects showing these lab abnormalities need to be followed up according to the 'DILI checklist' provided in the ISF. In case of clinical symptoms of hepatic injury (icterus, unexplained encephalopathy, unexplained coagulopathy, right upper quadrant abdominal pain, etc.) without lab results (ALT, AST, total bilirubin) available, the Investigator should make sure that these parameters are analysed, if necessary in an unscheduled blood test that needs to be sent to central laboratory. Should the results meet the criteria of hepatic injury alert, the procedures described in the DILI checklist should be followed.

#### • Severe or serious infections, opportunistic or mycobacterium tuberculosis infections

The opportunistic infections include pneumocystis jirovecii, Human Polyoma-1 virus disease including polyomavirus-associated nephropathy, Cytomegalie Virus, post-transplant lymphoproliferative disorder (Epstein-Barr-Virus), progressive multifocal leucoencephalopathy, bartonellosis (disseminated only), blastomycosis, toxoplasmosis, coccidioidomycosis, histoplasmosis, aspergillosis (invasive only), candidiasis (invasive


c41671420-01

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.

or pharyngeal), cryptococcosis, other invasive fungi (mucormycosis (zygomycosis, rhizopus, mucor, lichtheimia), scedosporium/ pseudallescheria boydii, fusarium), legionellosis, listeria monocytogenes (invasive only), tuberculosis, nocardiosis, nontuberculous mycobacterium, salmonellosis (invasive only), HBV reactivation, herpes simplex (invasive only), herpes zoster, strongyloides (hyperinfection syndrome and disseminated forms only), paracoccidioides, penicillium marneffei, sporothrix schenckii, cryptosporidium species (chronic only), microsporidiosis, leishmaniasis (visceral only), trypanosoma cruzi infection (Chagas' disease) (disseminated only), campylobacteriosis (invasive only), shigellosis (invasive only), vibriosis (invasive due to vibrio vulnificus), Hepatitis C progression [R17-2617 (15)].

#### • Vasculitis events

In this trial protocol vasculitis is defined as any event term included in the MedDRA SMQ Vasculitis (broad). This includes clinical and pathological features related to primary or secondary vasculitis syndromes and involving any type, size, and location of blood vessels.

According to ICH E3 (13), in addition to Deaths and serious adverse events, 'other significant' AEs need to be listed in the clinical trial report. These will be any non-serious adverse event that led to an action taken with study drug (e.g. discontinuation or dose reduced or interrupted).

An overall summary of adverse events will be presented.

The frequency of subjects with AEs will be summarised by treatment, primary system organ class (SOC) and preferred term (PT). Separate tables will be provided for subjects with serious AEs, for subjects with investigator-defined drug-related AEs, for subjects with investigator-defined drug-related serious adverse events and for subjects with AESIs. In addition, the frequency of subjects with AEs will be summarised by treatment, worst intensity, primary system organ class (SOC) and preferred term (PT).

The system organ classes will be sorted by default alphabetically, PTs will be sorted by descending frequency (within SOC).

In addition, frequencies of subjects with non-serious AEs that had an incidence of > 5% for at least one treatment will be summarised by treatment, primary SOC and PT.

#### 7.8.2 Laboratory data


The analyses of laboratory data will be descriptive in nature and will be based on BI standards as presented in "Handling, Display and Analysis of Laboratory Data" (14). Analyses will be based on normalised values, which means transforming to a standard unit and a standard reference range. The original values will be analysed if the transformation into standard unit is not possible for a parameter.

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.

Laboratory data will be analysed qualitatively via comparison of laboratory data to their reference ranges. Values outside the reference range as well as values defined as possibly clinically significant will be flagged in the data listings.

Clinically relevant findings in laboratory data will be reported as baseline conditions (at screening) or as AEs (during the trial) if judged clinically relevant by the investigator, and will be analysed as such.

It is the investigator's responsibility to decide whether a lab value is clinically significantly abnormal or not (at the RPM at the latest).

Descriptive statistics of laboratory data including change from baseline will be calculated by planned time point based on the worst value of the subject at that planned time point (or assigned to that planned time point).

#### 7.8.3 Vital signs

Descriptive statistics over time including change from baseline will be performed for vital signs (blood pressure and pulse rate). In the listing the change from baseline will also be displayed. In addition, the time profiles of median and (Min, Max) will be displayed graphically by treatment.

For post-dose measurements of vital signs, descriptive statistics will be calculated by planned time point based on the first value of the subject at that planned time point (or assigned to that planned time point).

Clinically relevant findings will be reported as baseline conditions (at screening) or as AEs (during the trial) if judged clinically relevant by the investigator, and will be analysed as such.

#### 7.8.4 ECG

Clinically relevant abnormal findings will be reported as adverse events. No separate listing or analysis of continuous ECG monitoring will be prepared.

#### 7.9 OTHER ANALYSIS

#### Physical examination


Physical examination findings will be reported as relevant medical history/baseline condition (i.e., a condition already existent before intake of trial drug) or as AE and will be summarised as such.

No separate listing or analysis of physical examination findings will be prepared.

# Boehringer Ingelheim TRIAL STATISTICAL ANALYSIS PLAN


1305-0024 c41671420-01

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.

# 7.9.1 Biomarker analyses

No biomarker analysis is planned.

# 7.9.2 PK/PD analyses

No PK/PD analysis is planned.

Date: 13 JUN 2023, Version 1.0 BI-VQD-12681\_50-415\_AD-01 (4.0)

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.

# 8. TIMEPOINT OF RELEASE OF TREATMENT INFORMATION

Not applicable due to open label fashion of the trial as described in the CTP section 4.1.5.

Date: 13 JUN 2023, Version 1.0 BI-VQD-12681\_50-415\_AD-01 (4.0)

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.

# 9. REFERENCES


| CPMP/ICH/363/96: "Statistical Principles for Clinical Trials", ICH Guideline Topic E9, Note For Guidance on Statistical Principles for Clinical Trials, current version. |
|---|
| <i>BI-VQD-12045_40-413:</i> "Identify and Manage Important Protocol Deviations (iPD)", current version, Group "Clinical Operations", KMED. |
| BI-KMED-BDS-TMP-0059: "iPD specification document (sdtm-dv-domain-specification)", template, current version, Group "Clinical Operations", KMED. |
| 001-MCS-50-415_RD-03: "Clinical Trial Analysis Decision Log (template)", current version, Group "Biostatistics & Data Sciences", KMED. |
| <i>BI-KMED-BDS-HTG-0035:</i> "Handling of Missing and Incomplete AE Dates", current version, Group "Biostatistics & Data Sciences" KMED. |
| <i>BI-KMED-TMCP-HTG-0025:</i> "Standards and processes for analyses performed within Clinical Pharmacokinetics/Pharmacodynamics", current version;, Group "Translational Medicine Clinical Pharmacology", KMED. |
| <i>BI-KMED-TMCP-MAN-0014:</i> "Noncompartmental Pharmacokinetic / Pharmacodynamic Analyses of Clinical Studies", current version, Group "Translational Medicine Clinical Pharmacology", KMED. |
| BI-KMED-BDS-HTG-0045: "Standards for Reporting of Clinical Trials and Project Summaries", current version, Group "Biostatistics & Data Sciences", KMED. |
| <i>BI-KMED-TMCP-OTH-0003</i> : "Graphs and Tables for Clinical Pharmacokinetics and Pharmacodynamic Noncompartmental Analyses", current version, Group "Translational Medicine Clinical Pharmacology", KMED. |
| <i>BI-KMED-TMCP-MAN-0010</i> : "Description of Analytical Transfer Files and PK/PD Data Files", current version, Group "Translational Medicine Clinical Pharmacology", KMED. |
| <i>BI-KMED-BDS-HTG-0041</i> : "Analysis and Presentation of Adverse Event Data from Clinical Trials – Display Template", current version, Group "Biostatistics & Data Sciences", KMED. |
| <i>BI-KMED-BDS-HTG-0066</i> : "Analysis and Presentation of AE data from clinical trials", current version, Group "Biostatistics & Data Sciences", KMED. |
| CPMP/ICH/137/95: "Structure and Content of Clinical Study Reports", ICH Guideline Topic E3; Note For Guidance on Structure and Content of Clinical Study Reports, current version, EMA webpage. |
| BI-KMED-BDS-HTG-0042: "Handling, Display and Analysis of Laboratory Data", current version, Group "Biostatistics & Data Sciences", KMED. |

# Boehringer Ingelheim TRIAL STATISTICAL ANALYSIS PLAN 1305-0024


c41671420-01

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.

15. *R17-2617:* Winthrop KL, Novosad SA, Baddley JW, Calabrese L, Chiller T, Polgreen P, et al. Opportunistic infections and biologic therapies in immune-mediated inflammatory diseases: consensus recommendations for infection reporting during clinical trials and postmarketing surveillance.

Ann Rheum Dis; 2015, 74; 2107-2116.

# Boehringer Ingelheim TRIAL STATISTICAL ANALYSIS PLAN 1305-0024


c41671420-01

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.

# 11. HISTORY TABLE

Table 11: 1 History table


| Version | Date<br>(DD-MMM-<br>YY) | Author | Sections changed | Brief description of change |
|---|---|---|---|---|
| 1.0 | 20-JUN-23 | | None | This is the final TSAP. |

BI-VQD-12681\_50-415\_AD-01 (4.0)